CLINICAL TRIAL: NCT01959464
Title: Sexual Absorption of Vaginal Progesterone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Carolinas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SAVP2013
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-07

CONDITIONS: Infertility; Pregnancy
Keywords: Assisted reproductive technology; Infertility; Progesterone; Vaginal gel; Luteal-phase support
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Initial assignment randomized, then crossed over to the other treatment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crinone vaginal progesterone gel (Experimental): Crinone is a bioadhesive vaginal gel containing micronized progesterone in an emulsion system containing a water swellable but insoluble polymer, polycarbophil. Crinone 8% is formulated to provide a long-acting vaginal retention, and is prescribed daily. Each applicator delivers 1.125 grams of Crinone gel containing 90 mg of progesterone. The reported time to maximum progesterone concentration is 6.8 +/- 3.3 hours with use of a single dose of Crinone 8%. Absorption half-life is approximately 25-50 hours and an elimination half-life of 5-20 minutes.
  On the evening of day 3, the female will insert the applicator into the vagina, administer the gel, and have intercourse within 1 hour of insertion of the cream.
  Interventions: Drug: Crinone vaginal progesterone gel
- Placebo vaginal gel (Placebo Comparator): The couple will be given a prefilled applicator containing either Crinone gel (progesterone) or placebo vaginal gel, data collection sheets and laboratory requisitions. On the evening of day 3, the female will insert the applicator into the vagina, administer the gel, and have intercourse within 1 hour of insertion of the cream.
  Interventions: Drug: Placebo vaginal gel

INTERVENTIONS:
Drug: Crinone vaginal progesterone gel — Crinone vaginal progesterone gel is inserted in the female vaginal using the pre-filled applicator.
  Arms: Crinone vaginal progesterone gel
Drug: Placebo vaginal gel — Placebo vaginal gel is inserted in the female vagina using the pre-filled applicator.
  Arms: Placebo vaginal gel

SUMMARY:
The purpose of this study is to determine if sexual intercourse lowers serum progesterone in women using vaginal progesterone gel (Crinone®), and increases serum progesterone in their male sexual partners. We hypothesize, based on previous estrogen studies done by our group, that intercourse will interfere with absorption of vaginal progesterone.

DETAILED DESCRIPTION:
The effects of intercourse on the absorption of vaginal progesterone for the female user and her sexual partner have not been studied. However, a previous study performed by our group found that intercourse lowered the absorption of vaginal estrogen cream in women, and men absorbed a small but statistically significant amount of estradiol during intercourse. Vaginal progesterone gel may be used by women for several clinical indications, and if intercourse alters the absorption and distribution of vaginal progesterone, clinical outcomes may be compromised. If intercourse lowers absorption, the efficacy of the treatment could be reduced. If intercourse enhances absorption, side effects may be increased. Also, if the male sexual partner absorbs vaginal progesterone, undesirable side effects may occur.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active 18-40 year old heterosexual couple
* Subject willing to take Mircette birth control pills for at least one cycle (one pack)
* Willing to have intercourse at the defined times (at least weekly within a 3 week interval, and draw blood within 10 hours of intercourse)
* IRB signed informed consent

Exclusion Criteria:

* Undiagnosed vaginal bleeding
* Contraindication to oral contraceptives
* Liver dysfunction or disease
* Known sensitivity to Crinone
* Known or suspected malignancy of the breast or genital organs
* History of or active thrombophlebitis or thromboembolic disorders
* Use of condoms during intercourse
* Male erectile or ejaculatory dysfunction

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Hurst, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
publication in manuscript

REFERENCES:
- [Background] Daya S, Gunby J. Luteal phase support in assisted reproduction cycles. Cochrane Database Syst Rev. 2004;(3):CD004830. doi: 10.1002/14651858.CD004830. PMID 15266541
- [Background] Yanushpolsky E, Hurwitz S, Greenberg L, Racowsky C, Hornstein M. Crinone vaginal gel is equally effective and better tolerated than intramuscular progesterone for luteal phase support in in vitro fertilization-embryo transfer cycles: a prospective randomized study. Fertil Steril. 2010 Dec;94(7):2596-9. doi: 10.1016/j.fertnstert.2010.02.033. Epub 2010 Mar 27. PMID 20347079
- [Background] Polyzos NP, Messini CI, Papanikolaou EG, Mauri D, Tzioras S, Badawy A, Messinis IE. Vaginal progesterone gel for luteal phase support in IVF/ICSI cycles: a meta-analysis. Fertil Steril. 2010 Nov;94(6):2083-7. doi: 10.1016/j.fertnstert.2009.12.058. Epub 2010 Feb 19. PMID 20171629
- [Background] Miles RA, Paulson RJ, Lobo RA, Press MF, Dahmoush L, Sauer MV. Pharmacokinetics and endometrial tissue levels of progesterone after administration by intramuscular and vaginal routes: a comparative study. Fertil Steril. 1994 Sep;62(3):485-90. doi: 10.1016/s0015-0282(16)56935-0. PMID 8062942
- [Background] De Ziegler D, Bulletti C, De Monstier B, Jaaskelainen AS. The first uterine pass effect. Ann N Y Acad Sci. 1997 Sep 26;828:291-9. doi: 10.1111/j.1749-6632.1997.tb48550.x. PMID 9329850
- [Background] Fonseca EB, Celik E, Parra M, Singh M, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Progesterone and the risk of preterm birth among women with a short cervix. N Engl J Med. 2007 Aug 2;357(5):462-9. doi: 10.1056/NEJMoa067815. PMID 17671254
- [Background] Cooper AJ. Progestogens in the treatment of male sex offenders: a review. Can J Psychiatry. 1986 Feb;31(1):73-9. doi: 10.1177/070674378603100116. PMID 2936441
- [Background] Cooper AJ, Sandhu S, Losztyn S, Cernovsky Z. A double-blind placebo controlled trial of medroxyprogesterone acetate and cyproterone acetate with seven pedophiles. Can J Psychiatry. 1992 Dec;37(10):687-93. doi: 10.1177/070674379203701003. PMID 1473073
- [Background] Money J. Treatment guidelines: antiandrogen and counseling of paraphilic sex offenders. J Sex Marital Ther. 1987 Fall;13(3):219-23. doi: 10.1080/00926238708403894. PMID 2959790
- [Background] Hurst BS, Jones AI, Elliot M, Marshburn PB, Matthews ML. Absorption of vaginal estrogen cream during sexual intercourse: a prospective, randomized, controlled trial. J Reprod Med. 2008 Jan;53(1):29-32. PMID 18251358
- [Background] Practice Committee of the American Society for Reproductive Medicine. Progesterone supplementation during the luteal phase and in early pregnancy in the treatment of infertility: an educational bulletin. Fertil Steril. 2008 Apr;89(4):789-92. doi: 10.1016/j.fertnstert.2008.02.012. PMID 18406835
- [Background] Practice Committee of the American Society for Reproductive Medicine. The clinical relevance of luteal phase deficiency: a committee opinion. Fertil Steril. 2012 Nov;98(5):1112-7. doi: 10.1016/j.fertnstert.2012.06.050. Epub 2012 Jul 20. PMID 22819186
- [Background] Watson Pharmaceuticals, Inc. Prescribing Information for Crinone. Available at: http://www.crinoneusa.com/professionals/Prescribing_Information.pdf. Retrieved April 22, 2011.
- [Derived] Merriam KS, Leake KA, Elliot M, Matthews ML, Usadi RS, Hurst BS. Sexual absorption of vaginal progesterone: a randomized control trial. Int J Endocrinol. 2015;2015:685281. doi: 10.1155/2015/685281. Epub 2015 Feb 3. PMID 25713585

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Women were enrolled into the study to receive the intervention; male partners also had blood samples taken
Groups:
- Placebo Vaginal Gel Then Crinone: The couple will be given a prefilled applicator containing placebo vaginal gel, data collection sheets and laboratory requisitions. On the evening of day 3, the female will insert the applicator into the vagina, administer the gel, and have intercourse within 1 hour of insertion of the cream. Then they will be crossed over to Crinone vaginal gel.
- Crinone Vaginal Progesterone Gel Then Placebo: Crinone is a bioadhesive vaginal gel containing micronized progesterone in an emulsion system containing a water swellable but insoluble polymer, polycarbophil. Crinone 8% is formulated to provide a long-acting vaginal retention, and is prescribed daily. Each applicator delivers 1.125 grams of Crinone gel containing 90 mg of progesterone. The reported time to maximum progesterone concentration is 6.8 +/- 3.3 hours with use of a single dose of Crinone 8%. Absorption half-life is approximately 25-50 hours and an elimination half-life of 5-20 minutes.
  On the evening of day 3, the female will insert the applicator into the vagina, administer the Crinone gel, and have intercourse within 1 hour of insertion of the cream. Then subject will cross over to placebo
Period: Overall Study
Arm/Group | Placebo Vaginal Gel Then Crinone | Crinone Vaginal Progesterone Gel Then Placebo
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Crinone Vaginal Progesterone Gel Then Placebo: Crinone is a bioadhesive vaginal gel containing micronized progesterone in an emulsion system containing a water swellable but insoluble polymer, polycarbophil. Crinone 8% is formulated to provide a long-acting vaginal retention, and is prescribed daily. Each applicator delivers 1.125 grams of Crinone gel containing 90 mg of progesterone. The reported time to maximum progesterone concentration is 6.8 +/- 3.3 hours with use of a single dose of Crinone 8%. Absorption half-life is approximately 25-50 hours and an elimination half-life of 5-20 minutes.
  On the evening of day 3, the female will insert the applicator into the vagina, administer the Crinone gel, and have intercourse within 1 hour of insertion of the cream. Then she will cross over to placebo.
- Placebo Vaginal Gel Then Crinone: The couple will be given a prefilled applicator containing placebo vaginal gel, data collection sheets and laboratory requisitions. On the evening of day 3, the female will insert the applicator into the vagina, administer the gel, and have intercourse within 1 hour of insertion of the cream. Then she will cross over to Crinone.
- Total: Total of all reporting groups
Arm/Group | Crinone Vaginal Progesterone Gel Then Placebo | Placebo Vaginal Gel Then Crinone | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Female Change in Progesterone
Description: The primary outcome variables will be: the change in serum progesterone levels increase after coitus in the female partner using vaginal progesterone gel compared to placebo
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: ng/ml
Groups:
- Crinone Vaginal Progesterone Gel: Crinone is a bioadhesive vaginal gel containing micronized progesterone in an emulsion system containing a water swellable but insoluble polymer, polycarbophil. Crinone 8% is formulated to provide a long-acting vaginal retention, and is prescribed daily. Each applicator delivers 1.125 grams of Crinone gel containing 90 mg of progesterone. The reported time to maximum progesterone concentration is 6.8 +/- 3.3 hours with use of a single dose of Crinone 8%. Absorption half-life is approximately 25-50 hours and an elimination half-life of 5-20 minutes.
  On the evening of day 3, the female will insert the applicator into the vagina, administer the gel, and have intercourse within 1 hour of insertion of the cream.
  Crinone vaginal progesterone gel: Crinone vaginal progesterone gel is inserted in the female vaginal using the pre-filled applicator.
Arm/Group | Placebo Vaginal Gel | Crinone Vaginal Progesterone Gel
Number analyzed (Participants) | 20 | 20
ng/ml | 0.8 [0.2 to 2.1] | 7.0 [3.5 to 11.9]

2. Secondary Outcome: Male Change in Progesterone
Description: The secondary outcome variable will be the change in serum progesterone levels after coitus in the male partner comparing vaginal progesterone gel and placebo.
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Placebo Vaginal Gel | Crinone Vaginal Progesterone Gel
Number analyzed (Participants) | 20 | 20
ng/ml | 0.54 [0.3 to 1.0] | 0.85 [0.2 to 1.8]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo Vaginal Gel | Crinone Vaginal Progesterone Gel
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No